CLINICAL TRIAL: NCT06519617
Title: Study on Optimization and Evaluation of Integrated Chinese and Western Medicine for Primary Sjogren's Syndrome Glandular Damage
Brief Title: Study on Optimization and Evaluation of Integrated Chinese and Western Medicine for pSS Glandular Damage
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Qingwen Tao (Other)
Responsible Party: Sponsor-Investigator, Qingwen Tao, chief physician of rheumatism department of Chinese-medicine, China-Japan Friendship Hospital
Organization: China-Japan Friendship Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-KY-173
Record Dates: First submitted 2024-07-13; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Primary Sjögren Syndrome
Keywords: randomized controlled trial
MeSH Terms: interventions — Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: The treatment group received an optimized program combining Chinese and Western medicine for pSS glandular injury, while the control group received a conventional program for pSS glandular injury.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional program group (Sham Comparator): Hydroxychloroquine Sulfate Tablets 200-400mg daily for 12 weeks.
  Interventions: Drug: Hydroxychloroquine Sulfate
- optimized program combining Chinese and Western medicine for pSS glandular damage (Active Comparator): The herbal prescription for patients eligible for qi and yin deficiency was 200 ml twice daily for 12 weeks.
  Interventions: Drug: Yi Qi Yang Yin Decoction

INTERVENTIONS:
Drug: Yi Qi Yang Yin Decoction — The Yi Qi Yang Yin Decoction (Dihuang 15g, Baihe 12g, Nanshashen 15g, celery Qinghao 10g, Malt 10g, Shengma 6g, Chaihu 6g) prescription for patients eligible for qi and yin deficiency was 200 ml twice daily for 12 weeks.
  Other Names: The treatment group
  Arms: optimized program combining Chinese and Western medicine for pSS glandular damage
Drug: Hydroxychloroquine Sulfate — Hydroxychloroquine Sulfate Tablets 200-400mg daily for 12 weeks.
  Other Names: the control group
  Arms: conventional program group

SUMMARY:
ChatGPT In a randomized controlled trial, 136 patients with primary Sjögren's syndrome (pSS) meeting the inclusion criteria were enrolled and randomly divided into two groups of 68 each. The treatment group received an optimized program combining Chinese and Western medicine for pSS glandular injury, while the control group received a conventional program for pSS glandular damage. The primary efficacy endpoint was the 12-week non-stimulated salivary flow rate (UWS) score. Secondary efficacy endpoints included the glandular damage Visual Analog Scale (VAS) scores, the European Sjögren's Syndrome Patient Reported Index (ESSPRI), among others. The treatment course lasted 12 weeks. The efficacy and safety of the optimized program for pSS glandular injury were evaluated by comparing within and between groups before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1. clinical diagnosis of pSS and qi and yin deficiency ; 2.Sign the informed consent form.

Exclusion Criteria:

* 1. pSS activity system damage (ESSDAI score ≥5); 2. Combined connective tissue diseases other than pSS; 3. Pregnant or lactating women; 4. severe cardiovascular and cerebrovascular diseases, liver and kidney failure, and severe malignant tumors; 5. taking psychotropic drugs; 6. assessed by the investigator to be ineligible for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2024-07-13 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
UWS score | 12 weeks after treatment
  unstimulated flow rate of saliva score. it is positive if the UWS ≤1.5 ml/15 min（or 0.1 ml/min). Higher scores(ml/min) mean a better outcome.

SECONDARY OUTCOMES:
VAS score | 12 weeks after treatment
  the glandular damage Visual Analog Scale score(dryness, fatigue and pain in the limbs). Patient self-assessed VAS scores ranged from 0 to 10. Higher scores mean a worse outcome.
ESSPRI | 12 weeks after treatment
  the European Sjögren's Syndrome Patient Reported Index, average of dryness, fatigue and pain in the limbs VAS scores. ESSPRI score varies from 0 to 10. Higher scores mean a worse outcome.
Schirmer test | 12 weeks after treatment
  Lacrimal secretion test. it is positive if the UWS ≤5 mm/5 min（or 1 mm/min). Higher scores(mm/min) mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Qingwem Tao, Study Chair — China-Japan Friendship Hospital
Locations (1):
- China-Japan friendship hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No